CLINICAL TRIAL: NCT00840827
Title: A Single-Arm, Open-Label Study of the Efficacy and Safety of Lenalidomide in Combination With Cyclosporine A in Patients With Red Blood Cell Transfusion-Dependent Myelodysplastic Syndromes
Brief Title: Efficacy and Safety of Lenalidomide in Combination With Cyclosporine A in Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0810010063
Record Dates: First submitted 2009-01-21; First posted 2009-02-10 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: stage (IPSS low and INT-1); RBC transfusion-dependent; non-del 5q MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients (Experimental): Lenalidomide 10mg po daily/ CSA 250mg orally twice daily
  Interventions: Drug: lenalidomide; Drug: cyclosporine A

INTERVENTIONS:
Drug: lenalidomide — Lenalidomide 10mg po daily
  Other Names: revlimid
Drug: cyclosporine A — CSA 250mg orally twice daily
  Other Names: Sandimmune

SUMMARY:
Lenalidomide has shown significant efficacy in the treatment of anemia associated with both 5q- and non 5q- MDS patients. The mechanism(s) of action of lenalidomide in MDS is still to be determined, but given the differences in response rates seen, it is probable that the mechanism is different for patients with 5q- disease compared to non 5q- patients. T-cell mediated activation of intramedullary apoptosis in patients with early MDS leading to impaired hematopoiesis has been well described. Immunomodulation with agents such as ATG, cyclosporine and thalidomide have demonstrated clear activity in some patients with MDS. Lenalidomide, among its many effects, is a potent immunomodulator, which may contribute to its ability to improve red blood cell counts in patients with MDS. It is possible that this effect could be augmented with the addition of cyclosporine A (CSA), in a similar manner to CSA effects in patients with other bone marrow failure syndromes such as aplastic anemia.

Subjects will be treated with lenalidomide 10 mg PO daily days 1-28 of a 28-day cycle. Cyclosporine A will be started on day 1 of cycle 2 (day 29) at a dose of 5 mg/kg per day given orally in 2 divided doses. Cyclosporine A levels will be assessed weekly and doses will be adjusted to maintain a serum trough level between 100-450 mg/ml. Patients will continue on therapy for minimum of 16 weeks unless toxicity occurs which precludes continuation on therapy, disease progression and/or patient withdrawal of consent. Patients not achieving response after completing 16 weeks of therapy will discontinue treatment. Patients achieving response will continue therapy until disease progression, unacceptable toxicity or loss of response.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age ≥ 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of low or intermediate-1 risk IPSS (MDS without an abnormality of chromosome 5 involving a deletion between bands q31 and q33. Red blood cell (RBC) transfusion-dependent anemia as having received ≥ 2 units of RBCs within 8 weeks on the first day of study treatment.
* ECOG performance status of ≤ 2 at study entry
* Laboratory test results within the following ranges:

  * Absolute neutrophil count (ANC) >500 x 109/L
  * Platelet count ≥ 50 x 109/L
  * Serum creatinine ≤ 2.0 mg/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) ≤ 2 x ULN
* Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must also agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take asprin (81 or 325 mg) daily as a prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide. Prior ≥ grade 3 NCI CTCAE (Version 3.0) allergic reaction/hypersensitivity.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type A, B, or C.
* Inability to aspirate bone marrow (dry tap).
* Proliferative (WBC ≥ 12,000/ul) CMML
* An abnormality of chromosome 5 involving a deletion between bands q31 and q 33.
* Any of the following lab abnormalities:

  * Absolute neutrophil count (ANC) <500 cells/mm3 (0.5 x 109/L)
  * Platelet count ≤ 50,000/mm3 (50 x 109/L)
  * Serum creatinine ≥ 2.5 mg/dL (221µmol/L)
  * Serum SGOT/AST or SGPT/ALT ≥ 2.0 x upper limit of normal (ULN)
  * Serum direct bilirubin ≥ 2.0 mg/dL (34µmol/L)
* Clinically significant anemia due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding (if a marrow aspirate is not evaluable for storage iron, transferring saturation must be ≥ 20% and serum ferritin not less than 50ng/mL).
* Use of hematopoietic growth factors within 7 days of the first day of study drug treatment.
* Chronic use (≥2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to ≥ 10mg/day of prednisone) within 28 days of the first study drug treatment.
* Use of experimental or standard drug (i.e chemotherapeutic, immunosuppressive, cytoprotective agents) for the treatment of MDS within 28 days of the first day of study drug
* Prior history of malignancy other than MDS except basal cell or squamous cell carcinoma in situ of the cervix or breast, unless the patient has been free of disease for ≥ 5 year.
* Myocardial infarction within 6 months prior to enrollment, or NYHA (New York Hospital Association) Class III or IV heart failure disease. History of active angina, congestive heart disease, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of uncontrolled ischemia and/or active conduction system abnormalities, or myocardial infarction within 6 months prior to enrollment, acute ischemia, or active conduction system abnormalities.
* Active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* History of thromboembolic event within the past 6 months prior to enrollment.
* Patients who have a hypersensitivity to Sandimmune® (cyclosporine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Feldman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Lenalidomide in Combination With Cyclosporine A (CSA) to Achieve Red Cell Transfusion Independence in Subjects With Low- or Intermediate-1 Risk IPSS MDS Without a Del (5q31-33) Cytogenetic Abnormality.
Description: Efficacy of lenalidomide + CSA will be evaluated as a function of red blood cell transfusion needs improvement (≥ 50% decrease in RBC transfusion requirements after 16 weeks of study treatment).
Time Frame: 16 weeks
Population: 6 patients were enrolled, the target enrollment was not met. Study was terminated by the PI and no statistical analysis was performed. None of the patients completed the 16 weeks of study treatment, therefore red blood cell transfusion could not be evaluated.
Arm/Group | All Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety of Lenalidomide in Combination With CSA in Subjects With Low- or Intermediate-1 Risk MDS Without a Del (5q31-33) Cytogenetic Abnormality by Type of Adverse Events.
Description: Safety will be evaluated by type of adverse events to lenalidomide in combination with CSA
Time Frame: 12 months
Population: 6 patients were enrolled, the target enrollment was not met. Study was terminated by the PI and no statistical analysis was performed. None of the patients completed the 12 months of study treatment, therefore the type of adverse events to lenalidomide in combination with CSA, could not be evaluated.
Arm/Group | All Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Tolerability of Lenalidomide in Combination With CSA in Subjects With Low- or Intermediate-1 Risk MDS Without a Del (5q31-33) Cytogenetic Abnormality by Frequency of Adverse Events.
Description: Tolerability will be evaluated by the frequency of adverse events to lenalidomide in combination with CSA
Time Frame: 12 months
Population: 6 patients were enrolled, the target enrollment was never met. Study was terminated by the PI and no statistical analysis was performed. None of the patients completed the 12 months of study treatment, therefore tolerability could not be evaluated.
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Primary Outcome: Efficacy of Lenalidomide in Combination With Cyclosporine A (CSA) to Achieve Red Cell Transfusion Independence in Subjects With Low- or Intermediate-1 Risk IPSS MDS Without a Del (5q31-33) Cytogenetic Abnormality.
Description: Efficacy of lenalidomide + CSA will be evaluated as a function of red blood cell transfusion independence.
Time Frame: 12 months
Population: 6 patients were enrolled, the target enrollment was not met. Study was terminated by the PI and no statistical analysis was performed. None of the patients completed the 12 months of study treatment, therefore red blood cell transfusion independence could not be evaluated.
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Primary Outcome: Efficacy of Lenalidomide in Combination With Cyclosporine A (CSA) to Achieve Red Cell Transfusion Independence in Subjects With Low- or Intermediate-1 Risk IPSS MDS Without a Del (5q31-33) Cytogenetic Abnormality by Hemoglobin Change.
Description: Efficacy of lenalidomide + CSA will be evaluated as a function of change of hemoglobin concentration from baseline to 12 months.
Time Frame: Baseline and 12 months
Population: 6 patients were enrolled, the target enrollment was not met. Study was terminated by the PI and no statistical analysis was performed. None of the patients completed the 12 months of study treatment, therefore the change of hemoglobin concentration from baseline to 12 weeks could not be evaluated.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Tolerability of Lenalidomide in Combination With CSA in Subjects With Low- or Intermediate-1 Risk MDS Without a Del (5q31-33) Cytogenetic Abnormality by Severity of Adverse Events.
Description: Tolerability will be evaluated by the severity of adverse events to lenalidomide in combination with CSA
Time Frame: 12 months
Population: as for outcome 3
Arm/Group | All Patients
Number analyzed (Participants) | 0

7. Secondary Outcome: Tolerability of Lenalidomide in Combination With CSA in Subjects With Low- or Intermediate-1 Risk MDS Without a Del (5q31-33) Cytogenetic Abnormality by the Relatedness of Adverse Events.
Description: Tolerability will be evaluated by the relatedness of adverse events to lenalidomide in combination with CSA
Time Frame: 12 months
Population: as for outcome 3
Arm/Group | All Patients
Number analyzed (Participants) | 0

8. Secondary Outcome: Safety of Lenalidomide in Combination With CSA in Subjects With Low- or Intermediate-1 Risk MDS Without a Del (5q31-33) Cytogenetic Abnormality by Frequency of Adverse Events.
Description: Safety will be evaluated by frequency of each type of adverse event to lenalidomide in combination with CSA
Time Frame: 12 months
Population: 6 patients were enrolled, the target enrollment was never met. Study was terminated by the PI and no statistical analysis was performed. None of the patients completed the 12 months of study treatment, therefore safety could not be evaluated.
Arm/Group | All Patients
Number analyzed (Participants) | 0

9. Secondary Outcome: Safety of Lenalidomide in Combination With CSA in Subjects With Low- or Intermediate-1 Risk MDS Without a Del (5q31-33) Cytogenetic Abnormality by Relatedness of Adverse Events to the Combination of Treatments.
Description: Safety will be evaluated by the relatedness of each type of adverse event to lenalidomide in combination with CSA
Time Frame: 12 months
Population: as for outcome 8
Arm/Group | All Patients
Number analyzed (Participants) | 0

10. Secondary Outcome: Safety of Lenalidomide in Combination With CSA in Subjects With Low- or Intermediate-1 Risk MDS Without a Del (5q31-33) Cytogenetic Abnormality by Severity of Adverse Events.
Description: Safety will be evaluated by the severity of each type of adverse event to lenalidomide in combination with CSA
Time Frame: 12 months
Population: as for outcome 8
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the 8th day of the study drug administration till discontinuation of study drug. An additional safety assessment was done 30 days (+/- 2 days) following the last dose of study drug.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=6)
Anemia (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 3
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Skin rash (Skin and subcutaneous tissue disorders) | 1
GERD (Gastrointestinal disorders) | 1
Intermittent Diarrhea (Gastrointestinal disorders) | 1
Nausea (General disorders) | 1
Lip tingling (General disorders) | 1
Decreased Vision (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No